CLINICAL TRIAL: NCT01012401
Title: Interactive Cancer Communication System (ICCS) in Lung Cancer: Evaluating Survival Benefits. Center of Excellence in Cancer Communication Research: Using Technology to Enhance Cancer Communication and Improve Clinical Outcomes
Brief Title: Evaluating an Interactive Cancer Communication System (ICCS) in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Hartford Hospital (Other); M.D. Anderson Cancer Center (Other); University of Illinois at Chicago (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M-2009-1223; 2P50CA095817-06 (NIH); XP08517 (Other: University of Wisconsin, Madison); NCI-2011-01004 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer, Stage IIIb or IV
Keywords: Lung cancer; Quality of life; Communication with physician
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHESS with Clinician Report + Internet access (Experimental): An Internet-based system, Comprehensive Health Enhancement Support System for Lung Cancer(CHESS-LC) integrates over 14 services to provide tailored cancer information, support, and interactive tools.
  Interventions: Other: CHESS website for lung cancer patient + internet access if needed
- Usual care with Internet access (Active Comparator): Control group patients will be given a list of URLs for 10-high quality lung cancer-related sites
  Interventions: Other: CHESS website for lung cancer patient + internet access if needed

INTERVENTIONS:
Other: CHESS website for lung cancer patient + internet access if needed — The Comprehensive Health Enhancement Support System (CHESS), a non-commercial, home-based system created by clinical, communication, and decision scientists at the University of Wisconsin, is distinguished by its quality, depth, and ease of use. It employs data on user health status to help users monitor their condition, guide them to tailored information and social support, make and implement important health decisions, and learn coping skills. Our tests and clinical trials demonstrate that an ICCS such as CHESS can be widely accepted and used, improve quality of life, information competence, and in some cases lead to more efficient use of health services. An Internet-based system, CHESS-LC integrates over 14 services to provide tailored cancer information, support, interactive tools, and communication with the clinical team.

SUMMARY:
This study will examine the potential for an Interactive Cancer Communication System (ICCS) to impact not only psychosocial outcomes such as quality of life but also length of survival in an advanced stage lung cancer population. Two hypotheses will be tested: the Comprehensive Health Enhancement Support System- Lung Cancer (CHESS- LC) will significantly improve patient quality of life and length of overall survival as compared to a usual care control group.

DETAILED DESCRIPTION:
The prognosis for Non-Small Cell Lung Cancer patients remains poor despite recent advances in anti-cancer therapies. A lung cancer diagnosis often inflicts fear, despair, and hopelessness on patients and loved ones. For lung cancer patients in particular, a population where palliation rather than cure is often the focus, interventions addressing communication about various types of suffering are crucial to quality of life (QOL). Our Center has done extensive research testing CHESS (Comprehensive Health Enhancement Support System), a non-commercial, web-based information and support system. The recent Clinician Integration Project tested the impact of CHESS versus an Internet only Control group on QOL for caregivers of advanced stage lung cancer patients. This study yielded an unanticipated finding that CHESS may have a survival benefit for patients as one year survival was significantly increased in the CHESS group (50%) compared to Internet (34.2%). As this project did not focus on patient outcomes, follow-up with a well-formulated study designed and powered to address specific hypotheses of the nature of this effect is critical. The proposed study will specifically test QOL and survival effects of CHESS on lung cancer patients. Using sites in Wisconsin, Connecticut,Houston, and Chicago, we will randomly assign 376 advanced lung cancer patients to two study arms: a patient control group receiving Usual Care (including access to a computer and Internet) and a group given access to the CHESS website. Patients may invite a caregiver to participate. Patients will be followed for 18 months or until patient death.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed with non-small cell lung cancer (Stage IIIA non surgical, IIIB or IV)
* All patients must be within 12 months of their primary lung cancer diagnosis or metastatic or recurrence disease.
* All patients must be at least 18 years of age,
* All patients must have an ECOG Performance Status rating of level 0, 1 or 2.
* If patients have brain metastases, they must be stable
* All patients must be under the care of a clinician who has consented to participate in the study.
* All patients must be able to speak and read English (educational attainment of at least 6th grade).
* All patients will be invited to have a caregiver also participate in the study, however this is not required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2014-05-15 (Actual); Study Completion 2014-05-15 (Actual)

PRIMARY OUTCOMES:
Compared to a Usual Care control, CHESS will significantly improve lung cancer patient Quality of Life. | 12-month intervention
Compared to a Usual Care control, CHESS will significantly improve patient influence length of survival of lung cancer patient. | 12-month intervention

SECONDARY OUTCOMES:
Examine the effects of CHESS use on self-determination theory (SDT) constructs. | 12 mos.
Examine the factors that moderate effect of CHESS use on self-determination theory (SDT) constructs. | 12 mos.
Examine whether these constructs mediate the effects of CHESS use on patient quality of life. | 12 mos.
Examine whether treatment participation mediates the effect patient quality of life has on survival. | 12 mos/

CONTACTS AND LOCATIONS:
Overall Officials: James Cleary, M.D., Principal Investigator — University of Wisconsin, Madison; Lori DuBenske, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- See also: Related Info — http://chess.wisc.edu/chess/projects/ICCS_Lung.aspx